CLINICAL TRIAL: NCT05161988
Title: Serum IL 26 as a Marker of Disease Activity in SLE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma alzahraa Mustafa Abdelbary Thabet, resident, Assiut University
Other Study IDs: SLE IL26
Record Dates: First submitted 2021-12-04; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: SLE

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assessment of serum Interleukin 26 level in SLE patients and compare it with healthy controls.

Association of serum interleukin 26 with SLE activity and severity.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic inflammatory disease characterized by diverse autoantibodies and varied clinical manifestations(mainly targeting the skin, kidneys, and brain). Autoantibodies directed against double-stranded (ds) DNA play a key role in the initiation and maintenance of inflammatory lesions in SLE(1).

Pathogenesis of SLE is mirrored by its complex aetiopathogenesis as genetic factors , environmental triggers (exposure to sunlight, drugs and infections, particularly with Epstein-Barr virus. . Causing secretion of inflammatory mediators , antibody and cytokines . But still pathological mechanisms of SLE are still not fully understood. (2) Immune system dysregulation such as incomplete clearance of apoptotic materials, hyperactivation of immune cells, overproduction of antibodies and abundant immune complex deposits are prominent in SLE (3) Clinical manifestations of SLE are Malar rash, Discoid rash ,Photosensitivity, Oral or nasopharyngeal ulcers, Pleurisy, Renal abnormalities, Immunologic abnormalities, Nonscarring alopecia, Synovitis, Hemolytic anemia, Leukopenia, Thrombocytopenia Proteinuria Seizures Psychosis Serositis and Arthritis (4) IL-26 is a 171-amino acid protein that belongs to the IL-10 family of cytokines, a family that includes IL-10, IL-19, IL-20, IL-22 and IL-24 . The IL-26 protein is encoded by the IL26 gene located on chromosome 12q15 between genes for interferon (IFN)-γ and IL-22 , and is conserved in several vertebrate species but not in mice and rats . The cytokine IL-26 was originally named AK155(5) IL-26 was initially identified as a pro-inflammatory cytokine , inducing the production of inflammatory cytokines by myeloid cells that are involved in the differentiation of naïve CD4+ T cells into Th17 cells (6) The involvement of IL 26 in numerous chronic auto inflammatory diseases and in two major pathogenic processes in SLE, namely the induction of IFN I and its production by Th 17 lymphocytes, makes the analysis of its role in SLE essential (7) Brilland et al., 2021 report that the levels of IL 26 are higher in SLE patients than healthy subjects and show a significant correlation with disease activity

ELIGIBILITY:
Inclusion Criteria:

* Adult SLE Patients who fulfilled the 2012 systemic lupus international collaborating clinics (SLICC) criteria

Exclusion Criteria:

* Individuals with other autoimmune diseases (rheumatoid arthritis dermatomyositis, scleroderma, mixed connective tissue disease).

Ages: 15 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Any patients fulfillef the critria o 2012 SLE international collaborating clinics and admition to Assiut University are participate in this study .
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-12-10 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of serum interleukin-26 level . | baseline
  Assessment of serum interleukin-26 level in SLE patients and compare it with the serum interleukin-26 level in healthy

SECONDARY OUTCOMES:
Association !! | baseline
  Association of serum interleukin 26 with SLE activity and severity.

REFERENCES:
- [Background] Knappe A, Hor S, Wittmann S, Fickenscher H. Induction of a novel cellular homolog of interleukin-10, AK155, by transformation of T lymphocytes with herpesvirus saimiri. J Virol. 2000 Apr;74(8):3881-7. doi: 10.1128/jvi.74.8.3881-3887.2000. PMID 10729163
- [Background] Maidhof W, Hilas O. Lupus: an overview of the disease and management options. P T. 2012 Apr;37(4):240-9. PMID 22593636
- [Background] Manson JJ, Rahman A. Systemic lupus erythematosus. Orphanet J Rare Dis. 2006 Mar 27;1:6. doi: 10.1186/1750-1172-1-6. PMID 16722594
- [Background] Roberts AL, Rizzolo D. Systemic lupus erythematosus: an update on treat-to-target. JAAPA. 2015 Sep;28(9):22-8. doi: 10.1097/01.JAA.0000470432.76823.93. PMID 26251978